CLINICAL TRIAL: NCT04839380
Title: An Open-Label, Single-Arm Study to Evaluate the Effect of Ruxolitinib 1.5% Cream on Itch in Adult Participants With Atopic Dermatitis
Brief Title: The Purpose of the Study is to Evaluate the Effect of Ruxolitinib Cream on Itch in Participants With Atopic Dermatitis
Acronym: SCRATCH-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-901
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
Keywords: ruxolitinib; Itch; Chronic Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — ruxolitinib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group : Ruxolitinib (Experimental): ruxolitinib cream 1.5% will be applied twice daily as a thin film.
  Interventions: Drug: ruxolitinib cream

INTERVENTIONS:
Drug: ruxolitinib cream — ruxolitinib cream 1.5% will be applied twice daily as a thin film
  Other Names: INCB018424

SUMMARY:
The purpose of the study is to evaluate the effect of ruxolitinib cream on itch in participants with Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Participant has clinically confirmed diagnosis of active AD for at least a 6-months.
* Participant has chronic pruritus related to AD for at least 3 months .
* Participant has an overall BSA (excluding palms, soles, scalp, genitals, and folds) affected by AD of 1%-20% on Day 1.
* Participant has an IGA score of at least 2 on Day 1.
* Participant has a single PP-NRS score ≥ 4 in the 24-hour period prior to the screening visit.
* Willingness to avoid pregnancy or fathering children.
* Participant must be willing to comply with all study procedures and restrictions including discontinuation of all current therapies for AD and pruritus (unless otherwise specified), and must be available for the duration of the study.

Exclusion Criteria:

* Female participnat who is breastfeeding, pregnant, or planning to become pregnant during the study.

Participant had significant flares or unstable course in AD.

* Participant has clinically infected AD or has used antibiotics (systemic or topical) for their infected AD within 2 weeks prior to the run-in period.
* Participant has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.
* Participant has any clinically significant medical condition or physical/laboratory/vital sign abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of study results.
* Participant has received treatment with JAK inhibitors (systemic or topical) within 4 weeks prior to the run-in period.
* Participant is unlikely, in the opinion of the investigator, to be compliant with study procedures and requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Innovaderm Research Inc., Montreal, Quebec
  - Innovoderm Research, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 study center in Canada.
Groups:
- Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for 28 days.
Period: Overall Study
Arm/Group | Ruxolitinib 1.5% Cream BID
Started | 49 (Safety Population: all enrolled participants who received at least 1 application of ruxolitinib 1.5% cream)
Intent-to-Treat Population | 46 (Participants who completed the Run-in Period and met all entry criteria.)
Completed | 44
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Dosed, but Did Not Complete Run-in Period | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (14.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Peak-Pruritus Numerical Rating Scale (PP-NRS) Score at Day 2 (24-hour Recall Period After First Application)
Description: The intensity of pruritus (itch) was recorded daily using the PP-NRS (24-hour recall period). Participants were asked to assign a numerical score representing their itch at the worst moment during the previous 24 hours on a scale of 0 to 10, with 0 being no itch and 10 being the worst itch imaginable. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the average of all non-missing PP-NRS scores reported during the 7-day run-in period.
Time Frame: Baseline; Day 2
Population: Modified Intent-to Treat (mITT) Population: all participants who had both a Baseline and at least 1 post-Baseline PP-NRS or modified PP-NRS (mPP-NRS) assessment within the treatment period. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
scores on a scale
  Baseline | 6.72 (1.363)
  Change from Baseline at Day 2: number analyzed (Participants) | 45
  Change from Baseline at Day 2 | -3.37 (1.847)

2. Secondary Outcome: Change From Baseline in the Modified Peak-Pruritus Numerical Rating Scale (mPP-NRS) Score (Current Itch Intensity) at 15 and 30 Minutes Postdose and at 1, 2, 4, 6, and 12 Hours Postdose on Day 1
Description: On Day 1, participants were asked to evaluate the current intensity of their itch at the time of assessment (i.e., prior to the morning study drug application, and 15 and 30 minutes and 1, 2, 4, 6, and 12 hours after the morning study drug application; the 12-hour evaluation occurred prior to the second daily study drug application) on a scale from 0 to 10, with 0 indicating no itch and 10 indicating the worst imaginable itch. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the last non-missing assessment before or on Day 1 and prior to the first application of study drug (including unscheduled assessments).
Time Frame: Baseline; Day 1 (15 and 30 minutes postdose; 1, 2, 4, 6, and 12 hours postdose)
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
scores on a scale
  Baseline | 6.4 (1.72)
  Change from Baseline at 15 minutes postdose | -2.3 (2.34)
  Change from Baseline at 30 minutes postdose | -3.0 (2.38)
  Change from Baseline at 1 hour postdose | -3.3 (2.45)
  Change from Baseline at 2 hours postdose | -3.8 (2.16)
  Change from Baseline at 4 hours postdose | -4.2 (2.12)
  Change from Baseline at 6 hours postdose | -4.2 (2.04)
  Change from Baseline at 12 hours postdose: number analyzed (Participants) | 43
  Change from Baseline at 12 hours postdose | -3.1 (2.00)

3. Secondary Outcome: Change From Baseline in the PP-NRS Score From Day 3 Through Day 29 (24-hour Recall Period After First Application)
Description: as for outcome 1
Time Frame: Baseline; Day 3 through Day 29
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
scores on a scale
  Baseline | 6.72 (1.363)
  Change from Baseline at Day 3: number analyzed (Participants) | 45
  Change from Baseline at Day 3 | -3.78 (1.775)
  Change from Baseline at Day 4: number analyzed (Participants) | 45
  Change from Baseline at Day 4 | -4.00 (1.760)
  Change from Baseline at Day 5 | -4.20 (1.875)
  Change from Baseline at Day 6: number analyzed (Participants) | 45
  Change from Baseline at Day 6 | -4.58 (1.935)
  Change from Baseline at Day 7 | -4.78 (1.755)
  Change from Baseline at Day 8: number analyzed (Participants) | 45
  Change from Baseline at Day 8 | -4.91 (1.832)
  Change from Baseline at Day 9: number analyzed (Participants) | 45
  Change from Baseline at Day 9 | -4.92 (1.890)
  Change from Baseline at Day 10: number analyzed (Participants) | 44
  Change from Baseline at Day 10 | -5.00 (1.762)
  Change from Baseline at Day 11: number analyzed (Participants) | 45
  Change from Baseline at Day 11 | -5.19 (1.606)
  Change from Baseline at Day 12: number analyzed (Participants) | 45
  Change from Baseline at Day 12 | -5.19 (1.722)
  Change from Baseline at Day 13: number analyzed (Participants) | 45
  Change from Baseline at Day 13 | -5.03 (1.907)
  Change from Baseline at Day 14: number analyzed (Participants) | 45
  Change from Baseline at Day 14 | -5.10 (1.745)
  Change from Baseline at Day 15: number analyzed (Participants) | 45
  Change from Baseline at Day 15 | -5.03 (1.805)
  Change from Baseline at Day 16: number analyzed (Participants) | 45
  Change from Baseline at Day 16 | -5.30 (1.680)
  Change from Baseline at Day 17: number analyzed (Participants) | 45
  Change from Baseline at Day 17 | -5.28 (1.510)
  Change from Baseline at Day 18: number analyzed (Participants) | 45
  Change from Baseline at Day 18 | -5.34 (1.826)
  Change from Baseline at Day 19: number analyzed (Participants) | 45
  Change from Baseline at Day 19 | -5.37 (1.739)
  Change from Baseline at Day 20: number analyzed (Participants) | 43
  Change from Baseline at Day 20 | -5.40 (1.759)
  Change from Baseline at Day 21: number analyzed (Participants) | 45
  Change from Baseline at Day 21 | -5.52 (1.692)
  Change from Baseline at Day 22: number analyzed (Participants) | 44
  Change from Baseline at Day 22 | -5.56 (1.726)
  Change from Baseline at Day 23: number analyzed (Participants) | 45
  Change from Baseline at Day 23 | -5.50 (1.598)
  Change from Baseline at Day 24: number analyzed (Participants) | 45
  Change from Baseline at Day 24 | -5.28 (1.773)
  Change from Baseline at Day 25: number analyzed (Participants) | 45
  Change from Baseline at Day 25 | -5.65 (1.629)
  Change from Baseline at Day 26: number analyzed (Participants) | 45
  Change from Baseline at Day 26 | -5.68 (1.585)
  Change from Baseline at Day 27: number analyzed (Participants) | 44
  Change from Baseline at Day 27 | -5.69 (1.689)
  Change from Baseline at Day 28: number analyzed (Participants) | 44
  Change from Baseline at Day 28 | -5.39 (1.845)
  Change from Baseline at Day 29: number analyzed (Participants) | 42
  Change from Baseline at Day 29 | -5.68 (1.595)

4. Secondary Outcome: Percentage of Participants Achieving at Least a 1-grade Decrease From Baseline in the mPP-NRS Score at 15 and 30 Minutes Postdose and at 1, 2, 4, 6, and 12 Hours Postdose on Day 1
Description: On Day 1, participants were asked to evaluate the current intensity of their itch at the time of assessment (i.e., prior to the morning study drug application, and 15 and 30 minutes and 1, 2, 4, 6, and 12 hours after the morning study drug application; the 12-hour evaluation occurred prior to the second daily study drug application) on a scale from 0 to 10, with 0 indicating no itch and 10 indicating the worst imaginable itch. Baseline was defined as the last non-missing assessment before or on Day 1 and prior to the first application of study drug (including unscheduled assessments). Confidence intervals were calculated using the Clopper-Pearson method.
Time Frame: Baseline; Day 1 (15 and 30 minutes postdose; 1, 2, 4, 6, and 12 hours postdose)
Population: mITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
percentage of participants
  15 minutes postdose | 82.6 [68.6 to 92.2]
  30 minutes postdose | 89.1 [76.4 to 96.4]
  1 hour postdose | 89.1 [76.4 to 96.4]
  2 hours postdose | 97.8 [88.5 to 99.9]
  4 hours postdose | 100.0 [92.3 to 100.0]
  6 hours postdose | 97.8 [88.5 to 99.9]
  12 hours postdose: number analyzed (Participants) | 43
  12 hours postdose | 90.7 [77.9 to 97.4]

5. Secondary Outcome: Percentage of Participants Achieving at Least a 1-grade Decrease From Baseline in the PP-NRS Score From Day 2 Through Day 29
Description: The intensity of pruritus (itch) was recorded daily using the PP-NRS (24-hour recall period). Participants were asked to assign a numerical score representing their itch at the worst moment during the previous 24 hours on a scale of 0 to 10, with 0 being no itch and 10 being the worst itch imaginable. Baseline was defined as the average of all non-missing PP-NRS scores reported during the 7-day run-in period.
Time Frame: Baseline; Day 2 through Day 29
Population: mITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
percentage of participants
  Day 2: number analyzed (Participants) | 45
  Day 2 | 93.3 [81.7 to 98.6]
  Day 3: number analyzed (Participants) | 45
  Day 3 | 95.6 [84.9 to 99.5]
  Day 4: number analyzed (Participants) | 45
  Day 4 | 97.8 [88.2 to 99.9]
  Day 5 | 97.8 [88.5 to 99.9]
  Day 6: number analyzed (Participants) | 45
  Day 6 | 97.8 [88.2 to 99.9]
  Day 7 | 97.8 [88.5 to 99.9]
  Day 8: number analyzed (Participants) | 45
  Day 8 | 97.8 [88.2 to 99.9]
  Day 9: number analyzed (Participants) | 45
  Day 9 | 97.8 [88.2 to 99.9]
  Day 10: number analyzed (Participants) | 44
  Day 10 | 97.7 [88.0 to 99.9]
  Day 11: number analyzed (Participants) | 45
  Day 11 | 100.0 [92.1 to 100.0]
  Day 12: number analyzed (Participants) | 45
  Day 12 | 100.0 [92.1 to 100.0]
  Day 13: number analyzed (Participants) | 45
  Day 13 | 100.0 [92.1 to 100.0]
  Day 14: number analyzed (Participants) | 45
  Day 14 | 97.8 [88.2 to 99.9]
  Day 15: number analyzed (Participants) | 45
  Day 15 | 100.0 [92.1 to 100.0]
  Day 16: number analyzed (Participants) | 45
  Day 16 | 100.0 [92.1 to 100.0]
  Day 17: number analyzed (Participants) | 45
  Day 17 | 100.0 [92.1 to 100.0]
  Day 18: number analyzed (Participants) | 45
  Day 18 | 100.0 [92.1 to 100.0]
  Day 19: number analyzed (Participants) | 45
  Day 19 | 97.8 [88.2 to 99.9]
  Day 20: number analyzed (Participants) | 43
  Day 20 | 97.7 [87.7 to 99.9]
  Day 21: number analyzed (Participants) | 45
  Day 21 | 100.0 [92.1 to 100.0]
  Day 22: number analyzed (Participants) | 44
  Day 22 | 100.0 [92.0 to 100.0]
  Day 23: number analyzed (Participants) | 45
  Day 23 | 100.0 [92.1 to 100.0]
  Day 24: number analyzed (Participants) | 45
  Day 24 | 97.8 [88.2 to 99.9]
  Day 25: number analyzed (Participants) | 45
  Day 25 | 100.0 [92.1 to 100.0]
  Day 26: number analyzed (Participants) | 45
  Day 26 | 100.0 [92.1 to 100.0]
  Day 27: number analyzed (Participants) | 44
  Day 27 | 100.0 [92.0 to 100.0]
  Day 28: number analyzed (Participants) | 44
  Day 28 | 97.7 [88.0 to 99.9]
  Day 29: number analyzed (Participants) | 42
  Day 29 | 100.0 [91.6 to 100.0]

6. Secondary Outcome: Percentage of Participants Achieving at Least a 2-grade Decrease From Baseline in the mPP-NRS Score at 15 and 30 Minutes Postdose and at 1, 2, 4, 6, and 12 Hours Postdose on Day 1
Description: On Day 1, participants were asked to evaluate the current intensity of their itch at the time of assessment (i.e., prior to the morning study drug application, and 15 and 30 minutes and 1, 2, 4, 6, and 12 hours after the morning study drug application; the 12-hour evaluation occurred prior to the second daily study drug application) on a scale from 0 to 10, with 0 indicating no itch and 10 indicating the worst imaginable itch. Baseline was defined as the last non-missing assessment before or on Day 1 and prior to the first application of study drug (including unscheduled assessments).
Time Frame: Baseline; Day 1 (15 and 30 minutes postdose; 1, 2, 4, 6, and 12 hours postdose)
Population: mITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
percentage of participants
  15 minutes postdose | 58.7 [43.2 to 73.0]
  30 minutes postdose | 67.4 [52.0 to 80.5]
  1 hour postdose | 71.7 [56.5 to 84.0]
  2 hours postdose | 91.3 [79.2 to 97.6]
  4 hours postdose | 95.7 [85.2 to 99.5]
  6 hours postdose | 93.5 [82.1 to 98.6]
  12 hours postdose: number analyzed (Participants) | 43
  12 hours postdose | 76.7 [61.4 to 88.2]

7. Secondary Outcome: Percentage of Participants Achieving at Least a 2-grade Decrease From Baseline in the PP-NRS Score From Day 2 Through Day 29
Description: as for outcome 5
Time Frame: Baseline; Day 2 through Day 29
Population: mITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
percentage of participants
  Day 2: number analyzed (Participants) | 45
  Day 2 | 71.1 [55.7 to 83.6]
  Day 3: number analyzed (Participants) | 45
  Day 3 | 82.2 [67.9 to 92.0]
  Day 4: number analyzed (Participants) | 45
  Day 4 | 84.4 [70.5 to 93.5]
  Day 5 | 87.0 [73.7 to 95.1]
  Day 6: number analyzed (Participants) | 45
  Day 6 | 91.1 [78.8 to 97.5]
  Day 7 | 95.7 [85.2 to 99.5]
  Day 8: number analyzed (Participants) | 45
  Day 8 | 93.3 [81.7 to 98.6]
  Day 9: number analyzed (Participants) | 45
  Day 9 | 95.6 [84.9 to 99.5]
  Day 10: number analyzed (Participants) | 44
  Day 10 | 95.5 [84.5 to 99.4]
  Day 11: number analyzed (Participants) | 45
  Day 11 | 97.8 [88.2 to 99.9]
  Day 12: number analyzed (Participants) | 45
  Day 12 | 97.8 [88.2 to 99.9]
  Day 13: number analyzed (Participants) | 45
  Day 13 | 95.6 [84.9 to 99.5]
  Day 14: number analyzed (Participants) | 45
  Day 14 | 97.8 [88.2 to 99.9]
  Day 15: number analyzed (Participants) | 45
  Day 15 | 97.8 [88.2 to 99.9]
  Day 16: number analyzed (Participants) | 45
  Day 16 | 100.0 [92.1 to 100.0]
  Day 17: number analyzed (Participants) | 45
  Day 17 | 97.8 [88.2 to 99.9]
  Day 18: number analyzed (Participants) | 45
  Day 18 | 95.6 [84.9 to 99.5]
  Day 19: number analyzed (Participants) | 45
  Day 19 | 95.6 [84.9 to 99.5]
  Day 20: number analyzed (Participants) | 43
  Day 20 | 97.7 [87.7 to 99.9]
  Day 21: number analyzed (Participants) | 45
  Day 21 | 97.8 [88.2 to 99.9]
  Day 22: number analyzed (Participants) | 44
  Day 22 | 97.7 [88.0 to 99.9]
  Day 23: number analyzed (Participants) | 45
  Day 23 | 100.0 [92.1 to 100.0]
  Day 24: number analyzed (Participants) | 45
  Day 24 | 95.6 [84.9 to 99.5]
  Day 25: number analyzed (Participants) | 45
  Day 25 | 100.0 [92.1 to 100.0]
  Day 26: number analyzed (Participants) | 45
  Day 26 | 100.0 [92.1 to 100.0]
  Day 27: number analyzed (Participants) | 44
  Day 27 | 97.7 [88.0 to 99.9]
  Day 28: number analyzed (Participants) | 44
  Day 28 | 95.5 [84.5 to 99.4]
  Day 29: number analyzed (Participants) | 42
  Day 29 | 97.6 [87.4 to 99.9]

8. Secondary Outcome: Time to Minimal Clinically Important Difference (MCID) for PP-NRS (≥2-grade Reduction in PP-NRS From Baseline )
Description: The MCID corresponds to an achievement of a ≥2-grade reduction in PP-NRS from Baseline. The time to MCID was defined as the time from the date (time) of the first dose to the date (time) of the first occurrence of MCID. Baseline was defined as the average of all non-missing PP-NRS scores reported during the 7-day run-in period.
Time Frame: from Baseline up to Day 29
Population: mITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
days | 1.6 (1.42)

9. Secondary Outcome: Time to MCID for mPP-NRS (≥2-grade Reduction in mPP-NRS From Baseline)
Description: The MCID corresponds to an achievement of a ≥2-grade reduction in mPP-NRS from Baseline. The time to MCID was defined as the time from the date (time) of the first dose to the date (time) of the first occurrence of MCID. Baseline was defined as the last non-missing assessment before or on Day 1 and prior to the first application of study drug (including unscheduled assessments).
Time Frame: Baseline; Day 1
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 45
hours | 0.817 (0.9788)

10. Secondary Outcome: Change From Baseline in Investigator Global Assessment (IGA) at Day 8, Day 15, and Day 29
Description: The IGA of the current state of the disease is a 5-point morphological assessment of overall disease severity. 0, clear: no erythema or induration/papulation, no oozing/crusting; there may be minor residual discoloration. 1, almost clear: there may be trace faint pink erythema with almost no induration/papulation and no oozing/crusting. 2, mild: there may be faint pink erythema with mild induration/papulation and no oozing/crusting. 3, moderate: there may be pink-red erythema with moderate induration/papulation, and there may be some oozing/crusting. 4, severe: there may be deep or bright red erythema with severe induration/papulation and with oozing/crusting.
Time Frame: Baseline; Days 8, 15, and 29
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
scores on a scale
  Baseline | 2.9 (0.31)
  Change from Baseline a Day 8: number analyzed (Participants) | 44
  Change from Baseline a Day 8 | -1.4 (0.73)
  Change from Baseline at Day 15: number analyzed (Participants) | 45
  Change from Baseline at Day 15 | -2.0 (0.87)
  Change from Baseline at Day 29: number analyzed (Participants) | 44
  Change from Baseline at Day 29 | -2.2 (0.90)

11. Secondary Outcome: Percentage of Participants Achieving Investigator Global Assessment-Treatment Success (IGA-TS) (Score of 0 or 1 in IGA With a ≥2-grade Reduction From Baseline) at Day 8, Day 15, and Day 29
Description: The IGA-TS is defined as an IGA score of 0 or 1 with a ≥2-grade reduction from Baseline. The IGA of the current state of the disease is a 5-point morphological assessment of overall disease severity. 0, clear: no erythema or induration/papulation, no oozing/crusting; there may be minor residual discoloration. 1, almost clear: there may be trace faint pink erythema with almost no induration/papulation and no oozing/crusting. 2, mild: there may be faint pink erythema with mild induration/papulation and no oozing/crusting. 3, moderate: there may be pink-red erythema with moderate induration/papulation, and there may be some oozing/crusting. 4, severe: there may be deep or bright red erythema with severe induration/papulation and with oozing/crusting.
Time Frame: Baseline; Days 8, 15, and 29
Population: mITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 46
percentage of participants
  Day 8: number analyzed (Participants) | 44
  Day 8 | 45.5 [30.4 to 61.2]
  Day 15: number analyzed (Participants) | 45
  Day 15 | 71.1 [55.7 to 83.6]
  Day 29: number analyzed (Participants) | 44
  Day 29 | 77.3 [62.2 to 88.5]

12. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. TEAEs were defined as any AEs with an onset date during or after the first study treatment dose.
Time Frame: up to Day 43
Population: Safety Analysis Set: all enrolled participants who received at least 1 application of ruxolitinib 1.5% cream.
Measure: Number; unit: participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 49
participants | 15

13. Secondary Outcome: Number of Participants With Any Grade 3 or Higher TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. TEAEs were defined as any AEs with an onset date during or after the first study treatment dose. The severity of AEs were assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to Day 43
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 49
participants | 0

ADVERSE EVENTS:
Time Frame: up to Day 43
Description: Treatment-emergent adverse events (TEAEs), defined as any adverse events with an onset date during or after the first study treatment dose, have been reported for all enrolled participants who received at least 1 application of ruxolitinib 1.5% cream (Safety Analysis Set).
Arm/Group | Ruxolitinib 1.5% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 15/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib 1.5% Cream BID (N=49)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
COVID-19 (Infections and infestations) | 3 (3)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Molluscum contagiosum (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT04839380/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT04839380/SAP_001.pdf